CLINICAL TRIAL: NCT01562236
Title: Gender-related Differences in Early Amplitude-integrated Electroencephalography in Newborns < 30 Weeks' Gestational Age and Their Correlation With Neurodevelopment Outcome at Three Years Corrected Age
Brief Title: Gender-specific aEEGs and Outcome in Preterms
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Monika Olischar, Ass Prof Dr, Medical University of Vienna
Other Study IDs: gender148
Record Dates: First submitted 2012-03-22; First posted 2012-03-23 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Gender Role Disorder, Male to Female Type

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Background and objectives: Male sex is a risk factor for poor neurodevelopmental outcome following preterm birth. The investigators aimed to investigate gender-related differences in amplitude-integrated electroencephalography (aEEG) and to correlate these findings with neurodevelopmental outcome.

Methods: Preterm infants born <30 weeks' gestational age between 2000 and 2002 were prospectively included. aEEGs obtained within the first two weeks of life were evaluated and classified according to background activity, sleep-wake cycling (SWC) and seizure activity. Outcome was assessed at three years.

ELIGIBILITY:
Inclusion Criteria:

* born<30 weeks gestational age
* who had aEEGs in first 2 weeks of life
* who were assessed for outcome at 3 years of age

Exclusion Criteria:

* born>30 weeks gestational age
* had no aEEGs in first 2 weeks of life
* lost for follow-up at 3 years

Ages: 24 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: preterms born < 30 weeks gestational age who had aEEG measurements within the first 2 weeks of life who had assessment of outcome at 3 years corrected age
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2000-01; Primary Completion 2002-12 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monika Olischar, MD, Principal Investigator — Neonatology
Locations (1):
- Medical University of Vienna, Vienna, Austria